CLINICAL TRIAL: NCT03678090
Title: The Safety and Efficacy of Fibrinolysis in Patients With an Indwelling Pleural Catheter for Multi-loculated Malignant Pleural Effusion: a Prospective Randomized Trial
Brief Title: The Safety and Efficacy of Fibrinolysis in Patients With an Indwelling Pleural Catheter for Multi-loculated Malignant Pleural Effusion.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Local IRB recommended IND exemption from FDA, study timeline not able to be met.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000024040
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Pleural Effusion; Cancer, Lung
MeSH Terms: conditions — Pleural Effusion; Lung Neoplasms | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tPA standard dosage (Active Comparator): Tissue Plasminogen Activator (tPA) dose of 10 to 25 mg.
  Interventions: Drug: tPA standard dosage
- tPA low dosage (Experimental): tPA dose of 2.5mg
  Interventions: Drug: tPA low dosage

INTERVENTIONS:
Drug: tPA standard dosage — Tissue plasminogen activator 25mg dosage
  Other Names: tissue plasminogen activator
  Arms: tPA standard dosage
Drug: tPA low dosage — Tissue plasminogen activator 2.5mg
  Other Names: tissue plasminogen activator
  Arms: tPA low dosage

SUMMARY:
The safety and efficacy of fibrinolysis in patients with an indwelling pleural catheter for multi-loculated malignant pleural effusion.

DETAILED DESCRIPTION:
Malignant pleural effusion (MPE) is a condition where fluid accumulates in the chest (pleural space) due to the presence of cancer. The malignancy may is usually metastatic from the lung, breast, or elsewhere and the presence of a MPE usually causes significant morbidity, particularly shortness of breath. Once a MPE develops, the patient's disease cannot be cured, but symptoms of dyspnea can be palliated.

Malignant effusions usually recur after thoracentesis, a procedure to remove the fluid. Upon recurrence, patients usually undergo placement of an indwelling pleural catheter (IPC). This is a small tube that drains fluid from inside the chest into a bottle to be discarded. It is very effective at treating shortness of breath and is safe.

On occasion, these catheters stop functioning, leading to an increase in the effusion again. This may be due to small amounts of blood or debris such as fibrin that clog the catheter, or it may be related to the pleural fluid becoming too thick to drain. Medication, namely tissue plasminogen activator (tPA), can be placed inside the catheter to promote drainage. With simple clogging, the tPA acts like "Draino." For fluid that has become too thick and pleural effusions that won't drain due to loculations, the tPA helps dissolve debris in the pleural fluid to promote drainage. Without this drainage, patients remain impaired due to shortness of breath related to the fluid.

tPA is effective at draining the fluid when debris has clogged the catheter or the pleural space. However, the exact dosing is unknown. For "simple" clogging, small doses may be used. When extensive loculations are present, large doses may be required to help the patient. Two retrospective studies have looked at very small doses of tPA placed through the IPC with the goal of breaking up the clogs in the catheter itself. These studies used between 2 and 5 mg of tPA.1,2 At Yale-New Haven Hospital, 25 mg has typically been used due to historical preference. It is unknown whether high doses of tPA improve its therapeutic efficacy.

The investigators hypothesize that higher dose fibrinolysis with 25mg of tPA (compared with 2.5 mg) will provide more effective clearance of fluid loculations, resulting in improved radiographic appearance and less shortness of breath without an increased risk of complications, such as bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Pleural Effusion MPE (either cytology proven or recurrent exudative pleural effusion in the context of histologically proven cancer)
* Presence of an indwelling pleural catheter (IPC)
* Nondraining IPC (defined as <50 mL of drainage on the past three drainage attempts) not responding to routine saline flush to assure patency
* Residual pleural fluid remaining on chest x-ray (CXR) or ultrasound
* Dyspnea deemed attributable to the effusion (i.e. symptomatic loculations), as assessed by the treating chest physician and using the modified Borg scale
* Presence of written informed consent from the patient or surrogate

Exclusion Criteria:

* Age <18
* Expected survival less than 14 days
* Known allergy or intolerance to tissue plasminogen activator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement in patient chest X-ray | up to 40 days
  Defined as change in percentage of hemithorax occupied by the pleural opacity on chest X-ray from the baseline chest X-ray to the X-ray at the end of the study protocol.
Improvement on the modified Borg dyspnea scale after tPA | up to 40 days
  Change in modified Borg dyspnea scale obtained at clinic visit where tPA is administered compared to modified Borg dyspnea scale obtained after post-tPA drainage.

SECONDARY OUTCOMES:
Time to recurrent loculation | up to 90 days
  In patients where tPA restores effective drainage, the time to and rate of patients who experience recurrent ineffective drainage due to loculation
Rate of pleurodesis | up to 90 days
  The rate of patients who are able to have the indwelling pleural catheter removed.
Improvements in dyspnea using the modified Borg scale | up to 40 days
  Change in modified Borg dyspnea scale obtained at initial clinic visit compared to scale at the end of the study protocol.

OTHER OUTCOMES:
Subgroup analysis of patients with trapped lung | up to 40 days
  We will also perform subgroup analysis by patients with trapped lung, stratification by primary tumor type, and stratification by the LENT score (a validated prognostic score for predicting mortality in patients with MPE).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Godfrey, MD, Principal Investigator — Yale University